CLINICAL TRIAL: NCT04087018
Title: A Phase 1b Study to Evaluate the Safety and Clinical Activity of AB122 in Biomarker-Selected Participants With Advanced Solid Tumors
Brief Title: Study to Evaluate Safety and Clinical Activity of AB122 in Biomarker Selected Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Strata Oncology (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB122CSP0002
Record Dates: First submitted 2019-08-29; First posted 2019-09-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TMB-H (Experimental): Participants with a tumor biomarker status of TMB-H will receive zimberelimab every 3 weeks.
  Interventions: Drug: zimberelimab
- Strata Immune Signature positive (Experimental): Participants with a tumor biomarker status Strata Immune Signature positive will receive zimberelimab every 3 weeks.
  Interventions: Drug: zimberelimab

INTERVENTIONS:
Drug: zimberelimab — zimberelimab is a fully human immunoglobulin G4 (IgG4) monoclonal antibody targeting human PD-1. Participants in each cohort will receive zimberelimab intravenously Q3W. Treatment will continue until progressive disease, unacceptable toxicity, withdrawal of consent, or other reasons for which investigational product discontinuation occurs.
  Other Names: AB122

SUMMARY:
This is a Phase 1b open-label study to evaluate the safety and clinical activity of zimberelimab (AB122) in biomarker-selected participants with advanced solid tumors.

DETAILED DESCRIPTION:
The activity of zimberelimab every 3 weeks (Q3W) will be evaluated in molecularly defined patient populations as described by the StrataNGS test (to be performed outside of this study protocol). Participants with any advanced tumor type will be stratified evenly by tumor biomarker status as follows: TMB-H or Strata Immune Signature positive. Each cohort may enroll approximately 40 participants. Following completion of and/or discontinuation from investigational product and follow-up, all participants will be followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* Male or female participants ≥ 18 years of age at the time of screening.
* Negative serum pregnancy test at screening and negative serum or urine pregnancy test every 3 months during the treatment period (women of childbearing potential only).
* Pathologically confirmed tumor that is metastatic, advanced, or recurrent with progression for which no alternative known to improve survival or curative therapy exists. Tumors must be TMB-H or Strata Immune Signature positive.
* Must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. The measurable lesion must be outside of a radiation field if the participant received prior radiation.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Prior chemotherapy or certain immune therapies or biologic agents must have been completed at least 4 weeks (28 days) before investigational product administration and all AEs have either returned to baseline or stabilized.
* Previously treated brain or meningeal metastases with no evidence of progression by magnetic resonance imaging (MRI) for at least 4 weeks (28 days) prior to the first dose.
* Immunosuppressive doses of systemic medications, such as corticosteroids or absorbed topical corticosteroids (doses > 10 mg/day prednisone or equivalent) must be discontinued at least 2 weeks (14 days) before investigational product administration. Physiologic doses of corticosteroids < 10 mg/day of prednisone or its equivalent may be permitted
* Prior surgery that required general anesthesia or other major surgery as defined by the Investigator must be completed at least 4 weeks before investigational product administration
* Negative tests for hepatitis B surface antigen, hepatitis C virus antibody (or hepatitis C qualitative ribonucleic acid [RNA; qualitative]), and human immunodeficiency virus (HIV)-1 and HIV-2 antibody at screening
* Adequate organ and marrow function

Exclusion Criteria:

* Use of any live attenuated vaccines against infectious diseases within 4 weeks (28 days) of initiation of investigational product.
* Underlying medical conditions that, in the Investigator's or Sponsor's opinion, will make the administration of investigational product hazardous or obscure the interpretation of toxicity determination or Adverse events (AEs).
* History of myocardial infarction within 6 months or history of arterial thromboembolic event within 3 months of the first dose of investigational agent.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the pre-screening or screening visit through 90 days after the last dose of investigational product.
* Any active or documented history of autoimmune disease or history of a syndrome that required systemic steroids or immunosuppressive medications.
* Any acute gastrointestinal symptoms at the time of screening or admission.
* Prior malignancy active within the previous year except for locally curable cancers that have been apparently cured.
* Prior treatment with an anti-PD-L1 or anti-PD-1 as monotherapy or in combination.
* Prior treatment with temozolomide.
* Use of other investigational drugs (drugs not marketed for any indication) within 28 days or at least 5 half-lives (whichever is longer) before investigational product administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Objective response Rate (ORR) | Approximately 12 months
  Based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Tumor assessments over time will be measured using RECIST v1.1

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) as Assessed by CTCAE v5.0 | From screening until 90 days after the last dose of investigational product or until initiation of a new systemic anticancer therapy, whichever occurs first, approximately 12 months
  Number of Participants Treated with zimberelimab with Treatment Emergent Adverse Events (TEAEs) as Assessed by CTCAE v5.0
Duration of response (DoR) | From the date of initiation of treatment until the date of first documented progression, through completion of the study, approximately 12 months
  The time from first documentation of disease response (CR or PR) until first documentation of progressive disease.
Time to response (TTR) | From the date of initiation of treatment until the date of first documented response, through completion of the study, approximately 12 months
  The time from treatment initiation to confirmed best overall response of CR or PR.
Disease control rate at 6 months (DCR6) | 6 Months
  Number of Participants with Complete Response, Partial Response, or Stable Disease for Greater Than 6 Months per RECIST v1.1
Progression-free survival at 6 (PFS6) | 6 Months
  The percentage of Participants Without Disease Progression per RECIST v1.1 and iRECIST at 6 months
Progression-free survival at 12 months (PFS12) | 12 Months
  The percentage of Participants Without Disease Progression per RECIST v1.1 and iRECIST at 12 months
Overall survival at 12 months (OS12) | 12 Months
  The percentage of participants who are alive at 12 months based on first dose to date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (9):
- United States (9):
  - Southern California Permanente Medical Group, Riverside, California
  - Kaiser Permanente (NorCal) - Roseville, Roseville, California
  - Christiana Care Health System - Helen F. Graham Cancer Center, Newark, Delaware
  - Kaiser Permanente Mid-Atlantic, Gaithersburg, Maryland
  - Metro MN CCOP, Saint Louis Park, Minnesota
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: AB122CSP0002 - Public website — https://trials.arcusbio.com/study/?id=AB122CSP0002